CLINICAL TRIAL: NCT02321592
Title: GHSG-AFM13 An Open-label, Randomized, Multicenter Phase II Trial With AFM13 in Patients With Relapsed or Refractory Hodgkin Lymphoma
Brief Title: GHSG-AFM13 An Open-label, Multicenter Phase II Trial With AFM13 in Patients With Relapsed or Refractory Hodgkin Lymphoma
Acronym: GHSG-AFM13
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Collaborators: Affimed GmbH (Industry); The Leukemia and Lymphoma Society (Other)
Responsible Party: Principal Investigator, Prof. Dr. Andreas Engert, Prof., University of Cologne
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Koeln-1754; 2014-004036-19 (EudraCT Number)
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Hodgkin Lymphoma
Keywords: Hodgkin Lymphoma; AFM13; Natural Killer Cells
MeSH Terms: conditions — Hodgkin Disease | interventions — AFM13

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A (Active Comparator): AFM13 is administered three times a week (e.g. monday-wednesday-friday) for 8 consecutive weeks.
  Arm A ist closed.
  Interventions: Drug: AFM13
- Arm B (Active Comparator): AFM13 is administered three times a week (e.g. monday-wednesday-friday) for 2 consecutive weeks followed by a weekly appication 6 consecutive weeks.
  Arm B is closed.
  Interventions: Drug: AFM13
- Arm C (Active Comparator): AFM13 is administered for five consecutive days a week as continuous infusion for 8 consecutive weeks
  Interventions: Drug: AFM13

INTERVENTIONS:
Drug: AFM13

SUMMARY:
The study is designed

* to demonstrate efficacy of AFM13 with an optimized treatment schedule
* to decide whether AFM13 warrants further investigation in a phase III clinical trial

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of classical HL reconfirmed by histopathology and relapsed or refractory disease after standard therapy including brentuximab vedotin and anti-PD1 or PD-L1 antibodies
* Age: 18 years or older (both genders)
* ECOG performance status ≤2
* Life expectancy >3 months
* Measurable site of disease with ≥ 1.5cm diameter which is evaluable by CT/MRI and FDG-avid by PET
* Completion of, if applicable, radiotherapy, chemotherapy, antibodies and immunoconjugates including brentuximab vedotin and/or another investigational drug which could interact with this trial not less than 4 weeks (or 5 half-lifes of the drug, whatever occurs later) prior to first dose of study drug
* Completion of, if applicable, an autologous stem cell transplantation (ASCT) at least 3 months prior tofirst dose of study drug
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care

Exclusion Criteria:

* Any significant diseases (other than HL) or clinically significant findings including psychiatric and behavioral problems, medical history and/or physical examination findings that would preclude the subject from participation in the study such as

  * unstable angina pectoris, symptomatic congestive heart failure (NYHA II, III, IV), myocardial infarction ≤ 6 months prior to first study drug, uncontrolled cardiac arrhythmia, cerebrovascular accidents ≤ 6 months before study drug start
  * severely impaired lung function as defined by spirometry (FEV1) and DLCO (diffusing capacity of the lung for carbon monoxide) that is 50% of the normal predicted value and/or O2 saturation that is 88% or less at rest on room air
  * Liver disease as indicated by AST >3 ULN (> 5 ULN if liver involvement is present)
  * any severe or uncontrolled other disease which might increase the risk associated with study participation or study drug administration and impair the ability to evaluate the patient or for the patient to complete the study
* Major organ dysfunction (except for HL-related reduced values e.g. in case of bone marrow or organ infiltration) as indicated by

  * Absolute Neutrophil Count (ANC) ≤1.5 x 109/l
  * Platelets <75 x 109/l
  * Hemoglobin level ≤9.0 g/dl (may be maintained by transfusions)
  * Total bilirubin >2 ULN (if >2 ULN direct bilirubin is required and should be ≤1.5 x ULN); Alkaline Phosphatase >3 ULN, AST or ALT ≥3 ULN (unless due to Hodgkin Lymphoma or diagnosed Gilbert´s Syndrome)
  * Blood creatinine level >2.0 mg/dl
* History of a previous malignancy ≤3 years prior to first dose of study drug except basal or squamous cell carcinoma of the skin, cervical carcinoma in situ or completely resected melanoma in stage TNMpT1
* Patients with a history of HIV seropositivity, chronic active hepatitis, or another uncontrolled active infection within 4 weeks prior to first dose of study drug
* Patients with evidence of current central nervous system (CNS) involvement
* Prior allogeneic stem cell transplantation (SCT)
* Patients receiving systemic corticosteroid treatment > 10 mg daily prednisone equivalents or other chronic systemic immunosuppressive agents within 2 weeks prior to first dose of study drug or during study treatment
* Major surgery within 4 weeks prior to first dose of study drug
* Known hypersensitivity to recombinant proteins or any excipient in the drug formulation
* General intolerance of any protocol medication including obligatory concomitant medication
* Pregnant or nursing women or women of childbearing potential not willing to use an effective form of contraception during participation in the study and at least 3 months thereafter. Male patients not willing to ensure that during the study and at least 3 months thereafter no fathering takes place
* Patient´s lack of accountability, inability to appreciate the nature, meaning and consequences of the trial and to formulate his/her own wishes correspondingly
* Patients unwilling to comply with the protocol
* Patients who have a relationship of dependence or employer-employee relationship to the sponsor or the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | at week 11

SECONDARY OUTCOMES:
Remission status based on CT/MRI and PET-CT | 3 weeks after end of treatment
Progression Free Survival (PFS) | 2 years
Overall Survival (OS) | 2 years
Adverse events (AEs) including acute treatment-associated toxicities | 2 years
Quality of Life (QoL)-score | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Engert, Prof., Principal Investigator — University Hospital of Cologne
Locations (1):
- 1st Department of Medicine, Cologne University Hospital, Cologne, Germany

REFERENCES:
- [Derived] Sasse S, Brockelmann PJ, Momotow J, Plutschow A, Huttmann A, Basara N, Koenecke C, Martin S, Bentz M, Grosse-Thie C, Thorspecken S, de Wit M, Kobe C, Dietlein M, Tresckow BV, Fuchs M, Borchmann P, Engert A. AFM13 in patients with relapsed or refractory classical Hodgkin lymphoma: final results of an open-label, randomized, multicenter phase II trial. Leuk Lymphoma. 2022 Aug;63(8):1871-1878. doi: 10.1080/10428194.2022.2095623. Epub 2022 Jul 18. PMID 35848865